CLINICAL TRIAL: NCT05236114
Title: TEMPUS GEMINI NSCLC STUDY: A Longitudinal Multi-Omic Biomarker Profiling Study of Patients With Non-Small Cell Lung Cancer (NSCLC)
Brief Title: GEMINI-NSCLC: NSCLC Biomarker Study
Status: Recruiting | Type: Observational
Sponsor: Tempus AI (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-CA-002
Record Dates: First submitted 2022-01-12; First posted 2022-02-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Cancer; Oncology; Observational; Genomic Profiling; Precision medicine; Non-Small Cell Lung Cancer; NSCLC; NGS; Biomarkers
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Cohort 1 will include patients with early-stage (Stages I-IIIB) who are candidates for treatment with curative intent, surgery with or without perioperative (neoadjuvant or adjuvant) therapy.
  Interventions: Other: Observation
- Cohort 2: Cohort 2 will include patients with stage IV disease receiving first line immunotherapy (as monotherapy or in combination with chemotherapy).
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — No intervention

SUMMARY:
GEMINI NSCLC Study is a non-interventional study that will be collecting clinical and molecular health information from patients with NSCLC who will receive longitudinal blood collection in addition to their standard of care therapy and disease surveillance with the goals of identifying the molecular evolution of lung cancer with standard of care therapy, and determining the utility of ctDNA dynamics to predict risk of recurrence and therapeutic outcomes.

ELIGIBILITY:
For Cohort 1 Inclusion, the participant has/is:

* A known or suspected NSCLC treated with curative intent -(surgery with or without perioperative (neoadjuvant or adjuvant) therapy).

  * Suspected NSCLC - Patients with a high index of suspicion for the diagnosis of NSCLC that is resectable may sign informed consent prior to undergoing diagnostic procedure at the discretion of the physician. NCCN Guidelines allow for clinical stage IA cancers to proceed directly to definitive surgery. Per NCCN Guidelines, if a preoperative tissue diagnosis has not been obtained, then an intraoperative diagnosis will be obtained. If a diagnosis of NSCLC is not confirmed and/or the tumor is not resectable, then the patient will be a screen failure.
* Undergone or planning to undergo a surgical resection - (Patients with stages I-IIIB who are resectable - per NCCN guidelines of resectability)
* Both patients who lack molecular abnormalities and those with identified molecular abnormalities may enroll. Choice of perioperative therapy is to follow SOC therapeutic guidelines for the participant's molecular and PD-L1 profile.
* 18 years old or older
* Willing and able to provide informed consent
* Willing to have additional blood samples collected during routine surveillance visits
* Must submit tumor sample representative of current disease

For Cohort 1 Exclusion, the participant has/is:

* Patients with superior sulcus tumors who are candidates for preoperative concurrent chemoradiation.
* Stage III locally advanced and unresectable patients who are candidates for chemoradiation followed by immunotherapy.
* It is expected that all patients on the cohort will be treated with a definitive surgical resection. Thus, clinical stage IIIB and IIIC patients who subsequently demonstrate pathologically confirmed N3 nodal disease or T4 N2 or 3 per any confirmatory procedure listed in NCCN guidelines for which definitive chemoradiotherapy rather than surgery is recommended per NCCN Guidelines are not eligible.
* Patients who receive primary radiation (in lieu of surgery if they are not surgical candidates).

For Cohort 2 Inclusion, the participant has/is:

* Histologically documented Stage IV NSCLC (de novo metastatic or relapse setting) not amenable to curative surgery or radiation therapy. Palliative radiation (for instance for impending bony fracture or to control pain) is allowed at any time during the protocol at the physician's discretion.
* Intended to receive first line immunotherapy (as monotherapy or in combination with chemotherapy). Patients who have had previous exposure to immunotherapy in the neoadjuvant or adjuvant setting are allowed to enroll as long as 12 months have elapsed since the prior exposure.

  * Patients in surveillance on Cohort 1 are eligible to roll over to Cohort 2 at the time of recurrence as long as they have had histologic confirmation of recurrence and have been off immunotherapy for 12 months or greater and meet all other inclusion/exclusion criteria.
* Tumors that lack activating EGFR mutations (e.g., exon 19 deletion or exon 21 L858R, exon 21 L861Q, exon 18 G719X, or exon 20 S768I mutation) and ALK fusions. Also, per NCCN Guideline recommended testing, tumors must also lack ROS1, BRAF, NTRK 1/2/3, METex14 skipping mutations, and RET for which there is available front-line targeted therapy. Only those patients with KRAS G12C mutations and ERBB2 (HER2) mutations with no contraindications to immunotherapy (PD-L1 1) for which there are no approved front-line targeted therapies and for whom immunotherapy would be the preferred front-line therapy are eligible.
* Patients may be enrolled with local molecular testing and those results will be provided.

  * Patients may be enrolled with local molecular testing and those results will be provided.
* 18 years and older
* Willing and able to provide informed consent
* Willing to have additional blood samples collected during routine surveillance visits
* Must submit tumor sample representative of current disease

Exclusion Criteria (both Cohorts):

* Patients without a known or suspected NSCLC diagnosis, or other disease processes such as sarcoidosis, lymphoma, or metastatic cancer from other sites.
* Not willing to have additional blood samples collected
* Patients with a secondary malignancy must have been both diagnosed > 2 years from the lung cancer of interest and have completed all therapy for that malignancy (including extended adjuvant therapy) > 2 years prior to diagnosis of the lung cancer of interest with the exception of the following:
* Patients with superficial basal cell carcinoma of low-risk histology per NCCN Guidelines (Low-risk histologic subtypes include nodular, superficial, and other non-aggressive growth patterns such as keratotic, infundibulocystic, and fibroepithelioma of Pinkus) and low-risk for recurrence per NCCN Guidelines (location on trunk or extremities, size < 2 cm, primary (not recurrent), with well-defined borders) can be included even if they are diagnosed < 2 years from the lung cancer of interest.
* Patients with superficial squamous cell carcinoma of low-risk pathology per NCCN Guidelines (verrucous, keratoacanthomatous) and low-risk for recurrence per NCCN Guidelines (located on trunk or extremities; 2 cm in size; primary lesion (vs. recurrent); well to moderately differentiated; < 2 mm thick and no invasion beyond subcutaneous fat; negative for perineural invasion; and negative for lymphatic or vascular involvement) can be included even if they are diagnosed < 2 years from the lung cancer of interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This protocol targets patients with Non-Small Cell Lung Cancer (NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Real-World Disease Free Survival (rwDFS) | 5 years
Real-World Overall Survival (rwOS) | 3 years

SECONDARY OUTCOMES:
Sensitivity, Specificity, PPV and NPV of MRD assay to predict recurrence at benchmark vs physician assessment of recurrence via conventional imaging every 6 months | 5 years
Sensitivity, Specificity, PPV and NPV of MRD assay to predict recurrence across longitudinal collections vs physician assessment of recurrence via conventional imaging every 6 months | 5 years
Real-World Disease Free Survival (rwDFS) stratified by ctDNA status at benchmark | 5 years
pCR rate stratified by ctDNA status | 5 years
Real-World Overall Survival (rwOS) stratified by ctDNA status at benchmark | 5 years
Positive percent agreement and negative percent agreement between plasma ctDNA vs tumor tissue at benchmark & longitudinal time points | 5 years
Real-World Overall Survival | 18 months
Real-World Progression-Free | 18 months
Treatment patterns | 18 months
Positive percent agreement and negative percent agreement between plasma ctDNA vs. tumor tissue at benchmark & longitudinal time points | 18 months

OTHER OUTCOMES:
Prevalence of genomic variants at landmark timepoints | 5 years
Compare ctDNA levels detected before and after biopsy | 5 years
Prevalence of genomic variants at landmark timepoints | 18 months
Identification of the emergence of genomic variants and tumor biologic subclones over time with early-stage and advanced stage lung cancer | 5 years
Identify genomic determinants of disease recurrence or progression. | 5 years
Define ctDNA status at clinically-meaningful timeframes: at completion of neoadjuvant therapy, at the completion of surgery, at the completion of adjuvant therapy, and 30 days post completion of all therapy. | 5 years
Correlate ctDNA clearance with the ability to obtain pCR | 5 years
Correlate ctDNA detection rate with stage of disease (stages I - III) | 5 years
Define ctDNA dynamics at specified surveillance timepoints and correlate with simultaneous imaging and clinical disease status | 5 years
Define PPV of ctDNA to predict recurrence | 5 years
Correlate ctDNA clearance (or lack of clearance) with rwPFS and rwOS. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Rhodes, MD, Principal Investigator — Tempus AI, Inc.
Locations (58):
- United States (58):
  - Alabama Oncology, Birmingham, Alabama
  - Mercy Clinic Oncology - Fort Smith, Fort Smith, Arkansas
  - MemorialCare, Fountain Valley, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - UCLA, Los Angeles, California
  - Eastern CT and Hematology and Oncology Associates, Norwich, Connecticut
  - Clermont Oncology Center, Clermont, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - Morehouse School of Medicine (MSM), Atlanta, Georgia
  - Piedmont Healthcare, Atlanta, Georgia
  - Hawaii Cancer Care, Honolulu, Hawaii
  - Southern Illinois Hospital Services, Carterville, Illinois
  - Cancer Care Specialists of Illinois, Decatur, Illinois
  - Northwestern University, Evanston, Illinois
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Community Health Network, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - The Center for Cancer and Blood Disorder, Bethesda, Maryland
  - Frederick Health Regional System, Frederick, Maryland
  - Mercy Clinic Oncology and Hematology - Joplin, Joplin, Missouri
  - Lake Regional Health System, Osage Beach, Missouri
  - Mercy Clinic Cancer and Hematology - Chub O'Reilly Cancer Center, Springfield, Missouri
  - Oncology Hematology Associates, Springfield, Missouri
  - Mercy Clinic Oncology and Hematology - Sindelar Cancer Center, St Louis, Missouri
  - Mercy Clinic Oncology and Hematology - David C. Pratt Cancer Center, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - OptumCare Cancer Care, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer Care Specialists Reno, Reno, Nevada
  - New Jersey Cancer Center, Belleville, New Jersey
  - New York Oncology Hematology, Albany, New York
  - Hematology Oncology Associates of Central New York, East Syracuse, New York
  - Cayuga Medical Center, Ithaca, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - White Plains Hospital, White Plains, New York
  - UNC, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Southeastern Medical Oncology Center (SMOC), Goldsboro, North Carolina
  - Aultman Hospital, Canton, Ohio
  - TriHealth Cancer Institute, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - OhioHealth Reseach Institute, Columbus, Ohio
  - Taylor Cancer Research Center, Maumee, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Mercy Clinic Oncology and Hematology - Coletta, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Oregon Oncology Specialists, Salem, Oregon
  - Cancer Care Associates of York, York, Pennsylvania
  - The Medical University of South Carolina, Charleston, South Carolina
  - Baptist Cancer Center, Memphis, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - PeaceHealth St. Joseph Medical Center-Bellingham, Bellingham, Washington
  - Cancer Care Northwest, Spokane Valley, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Gundersen Health System, La Crosse, Wisconsin

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Duma N, Santana-Davila R, Molina JR. Non-Small Cell Lung Cancer: Epidemiology, Screening, Diagnosis, and Treatment. Mayo Clin Proc. 2019 Aug;94(8):1623-1640. doi: 10.1016/j.mayocp.2019.01.013. PMID 31378236
- [Background] Chansky K, Sculier JP, Crowley JJ, Giroux D, Van Meerbeeck J, Goldstraw P; International Staging Committee and Participating Institutions. The International Association for the Study of Lung Cancer Staging Project: prognostic factors and pathologic TNM stage in surgically managed non-small cell lung cancer. J Thorac Oncol. 2009 Jul;4(7):792-801. doi: 10.1097/JTO.0b013e3181a7716e. PMID 19458556
- [Background] Pignon JP, Tribodet H, Scagliotti GV, Douillard JY, Shepherd FA, Stephens RJ, Dunant A, Torri V, Rosell R, Seymour L, Spiro SG, Rolland E, Fossati R, Aubert D, Ding K, Waller D, Le Chevalier T; LACE Collaborative Group. Lung adjuvant cisplatin evaluation: a pooled analysis by the LACE Collaborative Group. J Clin Oncol. 2008 Jul 20;26(21):3552-9. doi: 10.1200/JCO.2007.13.9030. Epub 2008 May 27. PMID 18506026
- [Background] Curran WJ Jr, Paulus R, Langer CJ, Komaki R, Lee JS, Hauser S, Movsas B, Wasserman T, Rosenthal SA, Gore E, Machtay M, Sause W, Cox JD. Sequential vs. concurrent chemoradiation for stage III non-small cell lung cancer: randomized phase III trial RTOG 9410. J Natl Cancer Inst. 2011 Oct 5;103(19):1452-60. doi: 10.1093/jnci/djr325. Epub 2011 Sep 8. PMID 21903745
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Faivre-Finn C, Reck M, Vansteenkiste J, Spigel DR, Wadsworth C, Melillo G, Taboada M, Dennis PA, Ozguroglu M; PACIFIC Investigators. Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC. N Engl J Med. 2018 Dec 13;379(24):2342-2350. doi: 10.1056/NEJMoa1809697. Epub 2018 Sep 25. PMID 30280658
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Jordan EJ, Kim HR, Arcila ME, Barron D, Chakravarty D, Gao J, Chang MT, Ni A, Kundra R, Jonsson P, Jayakumaran G, Gao SP, Johnsen HC, Hanrahan AJ, Zehir A, Rekhtman N, Ginsberg MS, Li BT, Yu HA, Paik PK, Drilon A, Hellmann MD, Reales DN, Benayed R, Rusch VW, Kris MG, Chaft JE, Baselga J, Taylor BS, Schultz N, Rudin CM, Hyman DM, Berger MF, Solit DB, Ladanyi M, Riely GJ. Prospective Comprehensive Molecular Characterization of Lung Adenocarcinomas for Efficient Patient Matching to Approved and Emerging Therapies. Cancer Discov. 2017 Jun;7(6):596-609. doi: 10.1158/2159-8290.CD-16-1337. Epub 2017 Mar 23. PMID 28336552
- [Background] Gobbini E, Swalduz A, Levra MG, Ortiz-Cuaran S, Toffart AC, Perol M, Moro-Sibilot D, Saintigny P. Implementing ctDNA Analysis in the Clinic: Challenges and Opportunities in Non-Small Cell Lung Cancer. Cancers (Basel). 2020 Oct 24;12(11):3112. doi: 10.3390/cancers12113112. PMID 33114393
- [Background] Aggarwal C, Thompson JC, Black TA, Katz SI, Fan R, Yee SS, Chien AL, Evans TL, Bauml JM, Alley EW, Ciunci CA, Berman AT, Cohen RB, Lieberman DB, Majmundar KS, Savitch SL, Morrissette JJD, Hwang WT, Elenitoba-Johnson KSJ, Langer CJ, Carpenter EL. Clinical Implications of Plasma-Based Genotyping With the Delivery of Personalized Therapy in Metastatic Non-Small Cell Lung Cancer. JAMA Oncol. 2019 Feb 1;5(2):173-180. doi: 10.1001/jamaoncol.2018.4305. PMID 30325992
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Lynch TJ, Bell DW, Sordella R, Gurubhagavatula S, Okimoto RA, Brannigan BW, Harris PL, Haserlat SM, Supko JG, Haluska FG, Louis DN, Christiani DC, Settleman J, Haber DA. Activating mutations in the epidermal growth factor receptor underlying responsiveness of non-small-cell lung cancer to gefitinib. N Engl J Med. 2004 May 20;350(21):2129-39. doi: 10.1056/NEJMoa040938. Epub 2004 Apr 29. PMID 15118073
- [Background] Maemondo M, Inoue A, Kobayashi K, Sugawara S, Oizumi S, Isobe H, Gemma A, Harada M, Yoshizawa H, Kinoshita I, Fujita Y, Okinaga S, Hirano H, Yoshimori K, Harada T, Ogura T, Ando M, Miyazawa H, Tanaka T, Saijo Y, Hagiwara K, Morita S, Nukiwa T; North-East Japan Study Group. Gefitinib or chemotherapy for non-small-cell lung cancer with mutated EGFR. N Engl J Med. 2010 Jun 24;362(25):2380-8. doi: 10.1056/NEJMoa0909530. PMID 20573926
- [Background] Ramalingam SS, Vansteenkiste J, Planchard D, Cho BC, Gray JE, Ohe Y, Zhou C, Reungwetwattana T, Cheng Y, Chewaskulyong B, Shah R, Cobo M, Lee KH, Cheema P, Tiseo M, John T, Lin MC, Imamura F, Kurata T, Todd A, Hodge R, Saggese M, Rukazenkov Y, Soria JC; FLAURA Investigators. Overall Survival with Osimertinib in Untreated, EGFR-Mutated Advanced NSCLC. N Engl J Med. 2020 Jan 2;382(1):41-50. doi: 10.1056/NEJMoa1913662. Epub 2019 Nov 21. PMID 31751012
- [Background] Soda M, Choi YL, Enomoto M, Takada S, Yamashita Y, Ishikawa S, Fujiwara S, Watanabe H, Kurashina K, Hatanaka H, Bando M, Ohno S, Ishikawa Y, Aburatani H, Niki T, Sohara Y, Sugiyama Y, Mano H. Identification of the transforming EML4-ALK fusion gene in non-small-cell lung cancer. Nature. 2007 Aug 2;448(7153):561-6. doi: 10.1038/nature05945. Epub 2007 Jul 11. PMID 17625570
- [Background] Solomon BJ, Mok T, Kim DW, Wu YL, Nakagawa K, Mekhail T, Felip E, Cappuzzo F, Paolini J, Usari T, Iyer S, Reisman A, Wilner KD, Tursi J, Blackhall F; PROFILE 1014 Investigators. First-line crizotinib versus chemotherapy in ALK-positive lung cancer. N Engl J Med. 2014 Dec 4;371(23):2167-77. doi: 10.1056/NEJMoa1408440. PMID 25470694
- [Background] Peters S, Camidge DR, Shaw AT, Gadgeel S, Ahn JS, Kim DW, Ou SI, Perol M, Dziadziuszko R, Rosell R, Zeaiter A, Mitry E, Golding S, Balas B, Noe J, Morcos PN, Mok T; ALEX Trial Investigators. Alectinib versus Crizotinib in Untreated ALK-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Aug 31;377(9):829-838. doi: 10.1056/NEJMoa1704795. Epub 2017 Jun 6. PMID 28586279
- [Background] Canon J, Rex K, Saiki AY, Mohr C, Cooke K, Bagal D, Gaida K, Holt T, Knutson CG, Koppada N, Lanman BA, Werner J, Rapaport AS, San Miguel T, Ortiz R, Osgood T, Sun JR, Zhu X, McCarter JD, Volak LP, Houk BE, Fakih MG, O'Neil BH, Price TJ, Falchook GS, Desai J, Kuo J, Govindan R, Hong DS, Ouyang W, Henary H, Arvedson T, Cee VJ, Lipford JR. The clinical KRAS(G12C) inhibitor AMG 510 drives anti-tumour immunity. Nature. 2019 Nov;575(7781):217-223. doi: 10.1038/s41586-019-1694-1. Epub 2019 Oct 30. PMID 31666701
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Gandhi L, Garassino MC. Pembrolizumab plus Chemotherapy in Lung Cancer. N Engl J Med. 2018 Sep 13;379(11):e18. doi: 10.1056/NEJMc1808567. No abstract available. PMID 30207917
- [Background] Addeo A, Passaro A, Malapelle U, Banna GL, Subbiah V, Friedlaender A. Immunotherapy in non-small cell lung cancer harbouring driver mutations. Cancer Treat Rev. 2021 May;96:102179. doi: 10.1016/j.ctrv.2021.102179. Epub 2021 Mar 19. No abstract available. PMID 33798954
- [Background] Siravegna G, Marsoni S, Siena S, Bardelli A. Integrating liquid biopsies into the management of cancer. Nat Rev Clin Oncol. 2017 Sep;14(9):531-548. doi: 10.1038/nrclinonc.2017.14. Epub 2017 Mar 2. PMID 28252003
- [Background] Crowley E, Di Nicolantonio F, Loupakis F, Bardelli A. Liquid biopsy: monitoring cancer-genetics in the blood. Nat Rev Clin Oncol. 2013 Aug;10(8):472-84. doi: 10.1038/nrclinonc.2013.110. Epub 2013 Jul 9. PMID 23836314
- [Background] Li BT, Janku F, Jung B, Hou C, Madwani K, Alden R, Razavi P, Reis-Filho JS, Shen R, Isbell JM, Blocker AW, Eattock N, Gnerre S, Satya RV, Xu H, Zhao C, Hall MP, Hu Y, Sehnert AJ, Brown D, Ladanyi M, Rudin CM, Hunkapiller N, Feeney N, Mills GB, Paweletz CP, Janne PA, Solit DB, Riely GJ, Aravanis A, Oxnard GR. Ultra-deep next-generation sequencing of plasma cell-free DNA in patients with advanced lung cancers: results from the Actionable Genome Consortium. Ann Oncol. 2019 Apr 1;30(4):597-603. doi: 10.1093/annonc/mdz046. PMID 30891595
- [Background] Leighl NB, Page RD, Raymond VM, Daniel DB, Divers SG, Reckamp KL, Villalona-Calero MA, Dix D, Odegaard JI, Lanman RB, Papadimitrakopoulou VA. Clinical Utility of Comprehensive Cell-free DNA Analysis to Identify Genomic Biomarkers in Patients with Newly Diagnosed Metastatic Non-small Cell Lung Cancer. Clin Cancer Res. 2019 Aug 1;25(15):4691-4700. doi: 10.1158/1078-0432.CCR-19-0624. Epub 2019 Apr 15. PMID 30988079
- [Background] Mack PC, Banks KC, Espenschied CR, Burich RA, Zill OA, Lee CE, Riess JW, Mortimer SA, Talasaz A, Lanman RB, Gandara DR. Spectrum of driver mutations and clinical impact of circulating tumor DNA analysis in non-small cell lung cancer: Analysis of over 8000 cases. Cancer. 2020 Jul 15;126(14):3219-3228. doi: 10.1002/cncr.32876. Epub 2020 May 4. PMID 32365229
- [Background] Ooki A, Maleki Z, Tsay JJ, Goparaju C, Brait M, Turaga N, Nam HS, Rom WN, Pass HI, Sidransky D, Guerrero-Preston R, Hoque MO. A Panel of Novel Detection and Prognostic Methylated DNA Markers in Primary Non-Small Cell Lung Cancer and Serum DNA. Clin Cancer Res. 2017 Nov 15;23(22):7141-7152. doi: 10.1158/1078-0432.CCR-17-1222. Epub 2017 Aug 29. PMID 28855354
- [Background] Reckamp KL, Melnikova VO, Karlovich C, Sequist LV, Camidge DR, Wakelee H, Perol M, Oxnard GR, Kosco K, Croucher P, Samuelsz E, Vibat CR, Guerrero S, Geis J, Berz D, Mann E, Matheny S, Rolfe L, Raponi M, Erlander MG, Gadgeel S. A Highly Sensitive and Quantitative Test Platform for Detection of NSCLC EGFR Mutations in Urine and Plasma. J Thorac Oncol. 2016 Oct;11(10):1690-700. doi: 10.1016/j.jtho.2016.05.035. Epub 2016 Jul 25. PMID 27468937
- [Background] Couraud S, Vaca-Paniagua F, Villar S, Oliver J, Schuster T, Blanche H, Girard N, Tredaniel J, Guilleminault L, Gervais R, Prim N, Vincent M, Margery J, Larive S, Foucher P, Duvert B, Vallee M, Le Calvez-Kelm F, McKay J, Missy P, Morin F, Zalcman G, Olivier M, Souquet PJ; BioCAST/IFCT-1002 investigators. Noninvasive diagnosis of actionable mutations by deep sequencing of circulating free DNA in lung cancer from never-smokers: a proof-of-concept study from BioCAST/IFCT-1002. Clin Cancer Res. 2014 Sep 1;20(17):4613-24. doi: 10.1158/1078-0432.CCR-13-3063. Epub 2014 Jul 10. PMID 25013125
- [Background] Kasi PM, Sawyer S, Guilford J, Munro M, Ellers S, Wulff J, Hook N, Krinshpun S, Koyen Malashevich A, Malhotra M, Rodriguez A, Moshkevich S, Grothey A, Kopetz S, Billings P, Aleshin A. BESPOKE study protocol: a multicentre, prospective observational study to evaluate the impact of circulating tumour DNA guided therapy on patients with colorectal cancer. BMJ Open. 2021 Sep 24;11(9):e047831. doi: 10.1136/bmjopen-2020-047831. PMID 34561256
- [Background] Hu Y, Ulrich BC, Supplee J, Kuang Y, Lizotte PH, Feeney NB, Guibert NM, Awad MM, Wong KK, Janne PA, Paweletz CP, Oxnard GR. False-Positive Plasma Genotyping Due to Clonal Hematopoiesis. Clin Cancer Res. 2018 Sep 15;24(18):4437-4443. doi: 10.1158/1078-0432.CCR-18-0143. Epub 2018 Mar 22. PMID 29567812
- [Background] Parikh AR, Van Seventer EE, Siravegna G, Hartwig AV, Jaimovich A, He Y, Kanter K, Fish MG, Fosbenner KD, Miao B, Phillips S, Carmichael JH, Sharma N, Jarnagin J, Baiev I, Shah YS, Fetter IJ, Shahzade HA, Allen JN, Blaszkowsky LS, Clark JW, Dubois JS, Franses JW, Giantonio BJ, Goyal L, Klempner SJ, Nipp RD, Roeland EJ, Ryan DP, Weekes CD, Wo JY, Hong TS, Bordeianou L, Ferrone CR, Qadan M, Kunitake H, Berger D, Ricciardi R, Cusack JC, Raymond VM, Talasaz A, Boland GM, Corcoran RB. Minimal Residual Disease Detection using a Plasma-only Circulating Tumor DNA Assay in Patients with Colorectal Cancer. Clin Cancer Res. 2021 Oct 15;27(20):5586-5594. doi: 10.1158/1078-0432.CCR-21-0410. Epub 2021 Apr 29. PMID 33926918
- [Background] Reinert T, Henriksen TV, Christensen E, Sharma S, Salari R, Sethi H, Knudsen M, Nordentoft I, Wu HT, Tin AS, Heilskov Rasmussen M, Vang S, Shchegrova S, Frydendahl Boll Johansen A, Srinivasan R, Assaf Z, Balcioglu M, Olson A, Dashner S, Hafez D, Navarro S, Goel S, Rabinowitz M, Billings P, Sigurjonsson S, Dyrskjot L, Swenerton R, Aleshin A, Laurberg S, Husted Madsen A, Kannerup AS, Stribolt K, Palmelund Krag S, Iversen LH, Gotschalck Sunesen K, Lin CJ, Zimmermann BG, Lindbjerg Andersen C. Analysis of Plasma Cell-Free DNA by Ultradeep Sequencing in Patients With Stages I to III Colorectal Cancer. JAMA Oncol. 2019 Aug 1;5(8):1124-1131. doi: 10.1001/jamaoncol.2019.0528. PMID 31070691
- [Background] Beaubier N, Tell R, Lau D, Parsons JR, Bush S, Perera J, Sorrells S, Baker T, Chang A, Michuda J, Iguartua C, MacNeil S, Shah K, Ellis P, Yeatts K, Mahon B, Taxter T, Bontrager M, Khan A, Huether R, Lefkofsky E, White KP. Clinical validation of the tempus xT next-generation targeted oncology sequencing assay. Oncotarget. 2019 Mar 22;10(24):2384-2396. doi: 10.18632/oncotarget.26797. eCollection 2019 Mar 22. PMID 31040929
- [Background] Beaubier N, Bontrager M, Huether R, Igartua C, Lau D, Tell R, Bobe AM, Bush S, Chang AL, Hoskinson DC, Khan AA, Kudalkar E, Leibowitz BD, Lozachmeur A, Michuda J, Parsons J, Perera JF, Salahudeen A, Shah KP, Taxter T, Zhu W, White KP. Integrated genomic profiling expands clinical options for patients with cancer. Nat Biotechnol. 2019 Nov;37(11):1351-1360. doi: 10.1038/s41587-019-0259-z. Epub 2019 Sep 30. PMID 31570899
- [Background] Finkle JD, Boulos H, Driessen TM, Lo C, Blidner RA, Hafez A, Khan AA, Lozac'hmeur A, McKinnon KE, Perera J, Zhu W, Dowlati A, White KP, Tell R, Beaubier N. Validation of a liquid biopsy assay with molecular and clinical profiling of circulating tumor DNA. NPJ Precis Oncol. 2021 Jul 2;5(1):63. doi: 10.1038/s41698-021-00202-2. PMID 34215841
- [Background] Lam V, Tran H, Vasquez M, et al. MA23.02 Circulating Tumor DNA Analysis with a Novel Variant Classifier for Recurrence Detection in Resected, Early-Stage Lung Cancer. Journal of Thoracic Oncology 2018;13(10):S438.
- [Background] Guardant Health, Inc. ORACLE: Observation of ResiduAl Cancer With Liquid Biopsy Evaluation. clinicaltrials.gov; 2021. Available from: https://clinicaltrials.gov/ct2/show/NCT05059444.
- [Background] Dafni U, Tsourti Z, Vervita K, Peters S. Immune checkpoint inhibitors, alone or in combination with chemotherapy, as first-line treatment for advanced non-small cell lung cancer. A systematic review and network meta-analysis. Lung Cancer. 2019 Aug;134:127-140. doi: 10.1016/j.lungcan.2019.05.029. Epub 2019 May 30. PMID 31319971
- [Background] Khongorzul P, Ling CJ, Khan FU, Ihsan AU, Zhang J. Antibody-Drug Conjugates: A Comprehensive Review. Mol Cancer Res. 2020 Jan;18(1):3-19. doi: 10.1158/1541-7786.MCR-19-0582. Epub 2019 Oct 28. PMID 31659006
- [Background] Brody R, Zhang Y, Ballas M, Siddiqui MK, Gupta P, Barker C, Midha A, Walker J. PD-L1 expression in advanced NSCLC: Insights into risk stratification and treatment selection from a systematic literature review. Lung Cancer. 2017 Oct;112:200-215. doi: 10.1016/j.lungcan.2017.08.005. Epub 2017 Aug 10. PMID 29191596
- [Background] Bratman SV, Yang SYC, Iafolla MAJ, Liu Z, Hansen AR, Bedard PL, Lheureux S, Spreafico A, Razak AA, Shchegrova S, Louie M, Billings P, Zimmermann B, Sethi H, Aleshin A, Torti D, Marsh K, Eagles J, Cirlan I, Hanna Y, Clouthier DL, Lien SC, Ohashi PS, Xu W, Siu LL, Pugh TJ. Personalized circulating tumor DNA analysis as a predictive biomarker in solid tumor patients treated with pembrolizumab. Nat Cancer. 2020 Sep;1(9):873-881. doi: 10.1038/s43018-020-0096-5. Epub 2020 Aug 3. PMID 35121950
- [Background] Litchfield K, Reading JL, Puttick C, Thakkar K, Abbosh C, Bentham R, Watkins TBK, Rosenthal R, Biswas D, Rowan A, Lim E, Al Bakir M, Turati V, Guerra-Assuncao JA, Conde L, Furness AJS, Saini SK, Hadrup SR, Herrero J, Lee SH, Van Loo P, Enver T, Larkin J, Hellmann MD, Turajlic S, Quezada SA, McGranahan N, Swanton C. Meta-analysis of tumor- and T cell-intrinsic mechanisms of sensitization to checkpoint inhibition. Cell. 2021 Feb 4;184(3):596-614.e14. doi: 10.1016/j.cell.2021.01.002. Epub 2021 Jan 27. PMID 33508232
- [Background] Fairfax BP, Taylor CA, Watson RA, Nassiri I, Danielli S, Fang H, Mahe EA, Cooper R, Woodcock V, Traill Z, Al-Mossawi MH, Knight JC, Klenerman P, Payne M, Middleton MR. Peripheral CD8+ T cell characteristics associated with durable responses to immune checkpoint blockade in patients with metastatic melanoma. Nat Med. 2020 Feb;26(2):193-199. doi: 10.1038/s41591-019-0734-6. Epub 2020 Feb 10. PMID 32042196
- [Background] Valpione S, Galvani E, Tweedy J, Mundra PA, Banyard A, Middlehurst P, Barry J, Mills S, Salih Z, Weightman J, Gupta A, Gremel G, Baenke F, Dhomen N, Lorigan PC, Marais R. Immune-awakening revealed by peripheral T cell dynamics after one cycle of immunotherapy. Nat Cancer. 2020 Feb;1(2):210-221. doi: 10.1038/s43018-019-0022-x. Epub 2020 Feb 10. PMID 32110781
- [Background] Nabet BY, Esfahani MS, Moding EJ, Hamilton EG, Chabon JJ, Rizvi H, Steen CB, Chaudhuri AA, Liu CL, Hui AB, Almanza D, Stehr H, Gojenola L, Bonilla RF, Jin MC, Jeon YJ, Tseng D, Liu C, Merghoub T, Neal JW, Wakelee HA, Padda SK, Ramchandran KJ, Das M, Plodkowski AJ, Yoo C, Chen EL, Ko RB, Newman AM, Hellmann MD, Alizadeh AA, Diehn M. Noninvasive Early Identification of Therapeutic Benefit from Immune Checkpoint Inhibition. Cell. 2020 Oct 15;183(2):363-376.e13. doi: 10.1016/j.cell.2020.09.001. Epub 2020 Oct 1. PMID 33007267
- [Background] Pellini B, Chaudhuri AA. Circulating Tumor DNA Minimal Residual Disease Detection of Non-Small-Cell Lung Cancer Treated With Curative Intent. J Clin Oncol. 2022 Feb 20;40(6):567-575. doi: 10.1200/JCO.21.01929. Epub 2022 Jan 5. PMID 34985936
- [Background] Kalvapudi S, Vedire Y, Yendamuri S, Barbi J. Neoadjuvant therapy in non-small cell lung cancer: basis, promise, and challenges. Front Oncol. 2023 Dec 8;13:1286104. doi: 10.3389/fonc.2023.1286104. eCollection 2023. PMID 38144524
- [Background] Wu YL, Tsuboi M, He J, John T, Grohe C, Majem M, Goldman JW, Laktionov K, Kim SW, Kato T, Vu HV, Lu S, Lee KY, Akewanlop C, Yu CJ, de Marinis F, Bonanno L, Domine M, Shepherd FA, Zeng L, Hodge R, Atasoy A, Rukazenkov Y, Herbst RS; ADAURA Investigators. Osimertinib in Resected EGFR-Mutated Non-Small-Cell Lung Cancer. N Engl J Med. 2020 Oct 29;383(18):1711-1723. doi: 10.1056/NEJMoa2027071. Epub 2020 Sep 19. PMID 32955177
- [Background] Tsuboi M, Herbst RS, John T, Kato T, Majem M, Grohe C, Wang J, Goldman JW, Lu S, Su WC, de Marinis F, Shepherd FA, Lee KH, Le NT, Dechaphunkul A, Kowalski D, Poole L, Bolanos A, Rukazenkov Y, Wu YL; ADAURA Investigators. Overall Survival with Osimertinib in Resected EGFR-Mutated NSCLC. N Engl J Med. 2023 Jul 13;389(2):137-147. doi: 10.1056/NEJMoa2304594. Epub 2023 Jun 4. PMID 37272535
- [Background] Felip E, Altorki N, Zhou C, Csoszi T, Vynnychenko I, Goloborodko O, Luft A, Akopov A, Martinez-Marti A, Kenmotsu H, Chen YM, Chella A, Sugawara S, Voong D, Wu F, Yi J, Deng Y, McCleland M, Bennett E, Gitlitz B, Wakelee H; IMpower010 Investigators. Adjuvant atezolizumab after adjuvant chemotherapy in resected stage IB-IIIA non-small-cell lung cancer (IMpower010): a randomised, multicentre, open-label, phase 3 trial. Lancet. 2021 Oct 9;398(10308):1344-1357. doi: 10.1016/S0140-6736(21)02098-5. Epub 2021 Sep 20. PMID 34555333
- [Background] Felip E, Altorki N, Zhou C, Vallieres E, Martinez-Marti A, Rittmeyer A, Chella A, Reck M, Goloborodko O, Huang M, Belleli R, McNally V, Srivastava MK, Bennett E, Gitlitz BJ, Wakelee HA. Overall survival with adjuvant atezolizumab after chemotherapy in resected stage II-IIIA non-small-cell lung cancer (IMpower010): a randomised, multicentre, open-label, phase III trial. Ann Oncol. 2023 Oct;34(10):907-919. doi: 10.1016/j.annonc.2023.07.001. Epub 2023 Jul 17. PMID 37467930
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Background] Forde PM, Spicer J, Lu S, Provencio M, Mitsudomi T, Awad MM, Felip E, Broderick SR, Brahmer JR, Swanson SJ, Kerr K, Wang C, Ciuleanu TE, Saylors GB, Tanaka F, Ito H, Chen KN, Liberman M, Vokes EE, Taube JM, Dorange C, Cai J, Fiore J, Jarkowski A, Balli D, Sausen M, Pandya D, Calvet CY, Girard N; CheckMate 816 Investigators. Neoadjuvant Nivolumab plus Chemotherapy in Resectable Lung Cancer. N Engl J Med. 2022 May 26;386(21):1973-1985. doi: 10.1056/NEJMoa2202170. Epub 2022 Apr 11. PMID 35403841
- [Background] Wakelee H, Liberman M, Kato T, Tsuboi M, Lee SH, Gao S, Chen KN, Dooms C, Majem M, Eigendorff E, Martinengo GL, Bylicki O, Rodriguez-Abreu D, Chaft JE, Novello S, Yang J, Keller SM, Samkari A, Spicer JD; KEYNOTE-671 Investigators. Perioperative Pembrolizumab for Early-Stage Non-Small-Cell Lung Cancer. N Engl J Med. 2023 Aug 10;389(6):491-503. doi: 10.1056/NEJMoa2302983. Epub 2023 Jun 3. PMID 37272513
- [Background] Spicer, J. D., et al. LBA56: Overall Survival in the KEYNOTE-671 study of Perioperative Pembrolizumab for Early-Stage Non-Small-Cell Lung Cancer (NSCLC). Annals of Oncology 2023 34(52):S1297.
- [Background] Sholl LM, Awad M, Basu Roy U, Beasley MB, Cartun RW, Hwang DM, Kalemkerian G, Lopez-Rios F, Mino-Kenudson M, Paintal A, Reid K, Ritterhouse L, Souter LA, Swanson PE, Ventura CB, Furtado LV. Programmed Death Ligand-1 and Tumor Mutation Burden Testing of Patients With Lung Cancer for Selection of Immune Checkpoint Inhibitor Therapies: Guideline From the College of American Pathologists, Association for Molecular Pathology, International Association for the Study of Lung Cancer, Pulmonary Pathology Society, and LUNGevity Foundation. Arch Pathol Lab Med. 2024 Jul 1;148(7):757-774. doi: 10.5858/arpa.2023-0536-CP. PMID 38625026
- [Background] Al Bakir M, Huebner A, Martinez-Ruiz C, Grigoriadis K, Watkins TBK, Pich O, Moore DA, Veeriah S, Ward S, Laycock J, Johnson D, Rowan A, Razaq M, Akther M, Naceur-Lombardelli C, Prymas P, Toncheva A, Hessey S, Dietzen M, Colliver E, Frankell AM, Bunkum A, Lim EL, Karasaki T, Abbosh C, Hiley CT, Hill MS, Cook DE, Wilson GA, Salgado R, Nye E, Stone RK, Fennell DA, Price G, Kerr KM, Naidu B, Middleton G, Summers Y, Lindsay CR, Blackhall FH, Cave J, Blyth KG, Nair A, Ahmed A, Taylor MN, Procter AJ, Falzon M, Lawrence D, Navani N, Thakrar RM, Janes SM, Papadatos-Pastos D, Forster MD, Lee SM, Ahmad T, Quezada SA, Peggs KS, Van Loo P, Dive C, Hackshaw A, Birkbak NJ, Zaccaria S; TRACERx Consortium; Jamal-Hanjani M, McGranahan N, Swanton C. The evolution of non-small cell lung cancer metastases in TRACERx. Nature. 2023 Apr;616(7957):534-542. doi: 10.1038/s41586-023-05729-x. Epub 2023 Apr 12. PMID 37046095
- [Background] Abbosh C, Frankell AM, Harrison T, Kisistok J, Garnett A, Johnson L, Veeriah S, Moreau M, Chesh A, Chaunzwa TL, Weiss J, Schroeder MR, Ward S, Grigoriadis K, Shahpurwalla A, Litchfield K, Puttick C, Biswas D, Karasaki T, Black JRM, Martinez-Ruiz C, Bakir MA, Pich O, Watkins TBK, Lim EL, Huebner A, Moore DA, Godin-Heymann N, L'Hernault A, Bye H, Odell A, Kalavakur P, Gomes F, Patel AJ, Manzano E, Hiley CT, Carey N, Riley J, Cook DE, Hodgson D, Stetson D, Barrett JC, Kortlever RM, Evan GI, Hackshaw A, Daber RD, Shaw JA, Aerts HJWL, Licon A, Stahl J, Jamal-Hanjani M; TRACERx Consortium; Birkbak NJ, McGranahan N, Swanton C. Tracking early lung cancer metastatic dissemination in TRACERx using ctDNA. Nature. 2023 Apr;616(7957):553-562. doi: 10.1038/s41586-023-05776-4. Epub 2023 Apr 13. PMID 37055640
- [Background] Wu YL, Dziadziuszko R, Ahn JS, Barlesi F, Nishio M, Lee DH, Lee JS, Zhong W, Horinouchi H, Mao W, Hochmair M, de Marinis F, Migliorino MR, Bondarenko I, Lu S, Wang Q, Ochi Lohmann T, Xu T, Cardona A, Ruf T, Noe J, Solomon BJ; ALINA Investigators. Alectinib in Resected ALK-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2024 Apr 11;390(14):1265-1276. doi: 10.1056/NEJMoa2310532. PMID 38598794
- [Background] O'Brien M, Paz-Ares L, Marreaud S, Dafni U, Oselin K, Havel L, Esteban E, Isla D, Martinez-Marti A, Faehling M, Tsuboi M, Lee JS, Nakagawa K, Yang J, Samkari A, Keller SM, Mauer M, Jha N, Stahel R, Besse B, Peters S; EORTC-1416-LCG/ETOP 8-15 - PEARLS/KEYNOTE-091 Investigators. Pembrolizumab versus placebo as adjuvant therapy for completely resected stage IB-IIIA non-small-cell lung cancer (PEARLS/KEYNOTE-091): an interim analysis of a randomised, triple-blind, phase 3 trial. Lancet Oncol. 2022 Oct;23(10):1274-1286. doi: 10.1016/S1470-2045(22)00518-6. Epub 2022 Sep 12. PMID 36108662